CLINICAL TRIAL: NCT00616694
Title: A Randomized Multicenter Parallel Group Study to Determine if Knowledge of Baseline Vertebral Fracture Prevalence (as Determined by Hologic IVA) and Bone Turnover Marker Determinations Improves Persistence With Actonel 5mg Daily Therapy in Subjects Receiving Chronic Glucocorticoid Therapy
Brief Title: Impact of Vertebral Fracture Knowledge on Persistence in Subjects Taking Glucocorticoid Therapy
Acronym: ACTIVATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR4003B_4027
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

INTERVENTIONS:
Drug: Actonel — Actonel 5 mg orally once daily (OD), calcium 500 mg + vitamin D 200 units twice daily (BID)
  Other Names: Risedronate Sodium

SUMMARY:
To evaluate the effect of subject knowledge of their disease status on persistence in subjects receiving Actonel 5 mg daily over a 12-month period for the prevention and treatment of GIO.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a variety of rheumatologic, pulmonary, and skin conditions.
* Subjects were to be on oral glucocorticoids with a mean daily dose of greater than or equal to 5.0 mg prednisone (or its equivalent) and were expected (although not required) to remain on a daily dose of greater than or equal to 5.0 mg prednisone (or its equivalent) for 12 months after the study started.
* Women must have been at least one year post-menopausal or surgically sterile.
* Subjects must have had evaluable BMD site at the lumbar spine (LS) and proximal femur.

Exclusion Criteria:

* Subject's unwillingness to take Vitamin D, calcium supplements or study medication
* A history of cancer: any history of cancer within the past 5 years. Relatively benign skin malignancies, such as basal cell carcinoma or squamous cell carcinoma, are not an exclusion if the subject has been in remission for at least 6 months prior to enrollment.
* A history of hyperparathyroidism, hyperthyroidism or osteomalacia or other metabolic bone disease within one year prior to enrollment
* History of alcohol or drug dependence within one year of enrollment
* A history of using any of the following medications within 6 months of starting study drug: Estrogen or estrogen-related drugs (tamoxifen, raloxifene, tibolone); low dose vaginal estrogen (estradiol < 0.2 mg/day, estropipate < 1.5 mg/day) will be allowed,Anabolic steroids,Parathyroid hormone
* A history of using any of the following medications within 1 month of starting study drugor for more than 1 month within 6 months prior to study entry: Calcitonin,Vitamin D supplements (>1000 IU per day),Calcitriol (>1.5mcg/week)
* A history of using any of the following medications within 6 months of starting study drug or for more than 14 days within 1 year prior to study entry: Any bisphosphonate,Fluoride (> 10 mg per day),Estrogen implant,Deflazacort
* Have received a depot injection of > 10,000 IU Vitamin D in the past 12 months
* Have a documented history of an abnormal or allergic reaction to bisphosphonates
* History of recurrent nephrolithiasis or a history of one episode of nephrolithiasis within 5years of study entry
* Severe renal impairment (creatinine clearance of <30 mL/min)
* Subjects on steroid therapy for transplantation
* Subjects on oral glucocorticoids for >8 weeks but <6 months at screening
* History of hypersensitivity to the investigational product or to drugs with similar chemical structures
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2002-07; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Determine whether subject knowledge of baseline vertebral fracture prevalence and awareness of results of bone turnover marker (BTM)determinations would result in an increase in persistence with Actonel 5 mg daily therapy | 12 months

SECONDARY OUTCOMES:
Evaluate relationship between prevalence of vertebral fractures and duration of prior steroid therapy, amount of prior steroid therapy, and diagnosis of disease for which steroids were used | 12 months
To evaluate the correlation between baseline vertebral fracture prevalence and subject persistence with Actonel 5 mg daily | 12 months
Evaluate influence of Actonel 5 mg on BTM determinations and bone mineral density(BMD) at study finish relative to baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States